CLINICAL TRIAL: NCT03306264
Title: A Phase 3, Randomized, Open-Label, Crossover Study of ASTX727 (Cedazuridine and Decitabine Fixed-Dose Combination) Versus IV Decitabine in Subjects With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), and Acute Myeloid Leukemia (AML)
Brief Title: Study of ASTX727 vs IV Decitabine in Participants With MDS, CMML, and AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-02; 2018-003395-12 (EudraCT Number)
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: MDS; CMML; decitabine; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; Decitabine; cedazuridine

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open-label, 2-period, 2-sequence crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MDS or CMML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 (Experimental): Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
  Interventions: Drug: ASTX727; Drug: Dacogen
- MDS or CMML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727 (Experimental): Participants with MDS or CMML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days) followed by ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
  Interventions: Drug: ASTX727; Drug: Dacogen
- AML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 (Experimental): Participants with AML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
  Interventions: Drug: ASTX727; Drug: Dacogen
- AML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727 (Experimental): Participants with AML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days) followed by ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
  Interventions: Drug: ASTX727; Drug: Dacogen

INTERVENTIONS:
Drug: ASTX727 — ASTX727 oral tablet
  Other Names: decitabine 35 mg + cedazuridine 100 mg
Drug: Dacogen — Decitabine 20 mg/m^2 one-hour IV infusion
  Other Names: decitabine

SUMMARY:
Multicenter PK study of ASTX727 versus IV decitabine. Adult participants who were candidates to receive IV decitabine were randomized 1:1 to receive the ASTX727 tablet Daily×5 in Cycle 1 followed by IV decitabine 20 mg/m^2 Daily×5 in Cycle 2, or the converse order. After completion of PK studies during the first 2 treatment cycles, participants continued to receive treatment with ASTX727 from Cycle 3 onward (in 28-day cycles) until disease progression, unacceptable toxicity, or the participants discontinued treatment or withdrew from the study.

DETAILED DESCRIPTION:
This Phase 3 study established PK equivalence of ASTX727 to IV decitabine in approximately 227 evaluable participants. Eligible participants were randomized to receive both study treatments: oral investigational drug ASTX727, and IV decitabine, as follows: participants were randomly assigned 1:1 to receive ASTX727 or IV decitabine in Cycle 1 and then cross over to the other therapy in Cycle 2.

In the ASTX727 cycle, participants received the ASTX727 tablet Daily×5. Serial PK measurements (blood draws) were done on Days 1, 2, and 5, along with pre-dose PK assessments on Days 1-5 and an assessment at 3 hours post-dose on Day 3. Participants were required to fast from food for 4 hours on days when receiving ASTX727: at least 2 hours before and 2 hours after dosing.

In the IV decitabine cycle, participants received a 1-hour infusion of IV decitabine 20 mg/m^2 Daily×5. Serial PK measurements were done on Days 1 and 5, along with pre-dose and 1-hour post-infusion assessments on Day 3.

In Cycles ≥3, participants received the ASTX727 tablet Daily×5 in 28-day cycles. (No PK assessments were done from Cycle 3 onward.)

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure; specifically able to comply with the PK assessment schedule during the first 2 treatment cycles.
2. Men or women ≥18 years who are candidates to receive IV decitabine according to FDA or European Medicines Agency (EMA) approved indications:

   1. In North America: Participants with MDS previously treated or untreated with de novo or secondary MDS, including all French-American-British subtypes (refractory anemia, refractory anemia with ringed sideroblasts, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, and chronic myelomonocytic leukemia [CMML]), and subjects with MDS International Prognostic Scoring System (IPSS) int-1, -2, or high-risk MDS.
   2. In Europe: Participants with de novo or secondary AML, as defined by the World Health Organization (WHO) criteria, who are not candidates for standard induction chemotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Adequate organ function defined as follows:

   1. Hepatic: Total or direct bilirubin ≤2 × upper limit of normal (ULN); aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) ≤2.5 × ULN.
   2. Renal: serum creatinine ≤1.5 × ULN or calculated creatinine clearance or glomerular filtration rate >50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
5. No major surgery within 30 days of first study treatment.
6. Life expectancy of at least 3 months.
7. Women of child-bearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of non-childbearing potential are those who have had a hysterectomy or bilateral oophorectomy, or who have completed menopause, defined as no menses for at least 1 year AND either age ≥65 years or follicle-stimulating hormone levels in the menopausal range.
8. Subjects and their partners with reproductive potential must agree to use effective contraceptive measures during the study and for 3 months after the last dose of study treatment. Effective contraception includes methods such as oral contraceptives or double-barrier method (eg, use of a condom AND diaphragm, with spermicide).

Exclusion Criteria:

1. Prior treatment with more than 1 cycle of azacitidine or decitabine. Prior cytotoxic chemotherapy for AML except for hydroxyurea to control high white blood cell (WBC) counts.
2. Hospitalization for more than 2 days for documented febrile neutropenia, pneumonia, sepsis, or systemic infection in the 30 days before screening.
3. Treatment with any investigational drug or therapy within 2 weeks of study treatment, or 5 half-lives, whichever is longer, before the first dose of study treatment, or ongoing clinically significant adverse events (AEs) from previous treatment.
4. Cytotoxic chemotherapy or prior azacitidine or decitabine within 4 weeks of first dose of study treatment.
5. Concurrent MDS therapies, including lenalidomide, erythropoietin, cyclosporine/tacrolimus, granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor, etc. (Prior treatment with these agents is permitted, provided that completion is at least 1 week before the first dose of study treatment.)
6. Poor medical risk because of other conditions such as uncontrolled systemic diseases, active uncontrolled infections, or comorbidities that may put the patient at risk of not being able to complete at least 2 cycles of treatment.
7. Known significant mental illness or other condition, such as active alcohol or other substance abuse or addiction, that in the opinion of the investigator predisposes the subject to high risk of noncompliance with the protocol.
8. Rapidly progressive or highly proliferative disease (total white blood cell count of >15 × 10^9/L) or other criteria that render the subject at high risk of requiring intensive cytotoxic chemotherapy within the next 3 months.
9. Life-threatening illness or severe organ system dysfunction, such as uncontrolled congestive heart failure or chronic obstructive pulmonary disease, or other reasons including laboratory abnormalities, which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ASTX727, or compromise completion of the study or integrity of the study outcomes.
10. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, prostate cancer or breast cancer under control with hormone therapy, or other cancer from which the subject has been disease free for at least 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (39):
  - Pinnacle Research Group, Anniston, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Compassionate Cancer Care Research Group, Fountain Valley, California
  - University of Southern California, Los Angeles, California
  - Yale, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Boca Raton Clinical Research, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai, Miami Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Regional Cancer Care Associates, Bethesda, Maryland
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hackensack, Hackensack, New Jersey
  - Roswell Park, Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore, The Bronx, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - West Penn Allegheny Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Vanderbilt, Nashville, Tennessee
  - Baylor Scott & White University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Austria (3):
  - Uniklinikum Salzburg, Salzburg
  - General Hospital Hietzing, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen Elizabeth II (QEII) Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Hospital & Cancer Center, Hamilton, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Center - University Health Network, Toronto, Ontario
  - Centre Intégré Universitaire de Santé et de Services Sociaux (CIUSSS) de l'Est-de-l'Ile-de-Montréal - Hôpital Maisonneuve Rosemont, Montreal, Quebec
- Czechia (3):
  - FN Ostrava, Ostrava, Poruba
  - University Hospital Brno, Brno
  - Fakultni Nemocnice Kralovske Vinohrady FNKV, Prague, Česká Republika
- France (2):
  - Centre de lutte contre le Cancer Leon Berard, Lyon, Rhone
  - Hospital Emile Muller, Mulhouse
- Germany (7):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden
  - Philipps-Universität Marburg, Klinik für Innere medizin, Hämatologie, Onkologie und Immunologie, Marburg, Hesse
  - UNIVERSITTSKLINIKUM Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Oberärztin für Innere Medizin, Hämato-/Onkologie und Palliativmedizin, Düsseldorf
  - University Hospital Halle, Halle
  - University of Leipzig, Leisnig
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei KAposi Mor Oktato Korhaz, Kaposvár
  - University of Pecs, 1st Department of Internal Medicine, Pécs
  - University of Szeged, Szeged
- Italy (6):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS C Granda OM Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità Novara, Novara
  - Ospedale S. Eugenio, Rome
  - ULSS 8 Vicenza - Ospedale San Bortolo di Vicenza, Vicenza
- Spain (11):
  - Hospital U. Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clinica Universitaria Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universitaria Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari I Politècnic La Fe, Valencia
- United Kingdom (2):
  - Oxford University Hopsitals NHS Trust, Oxford, Oxfordshire
  - The Christie NHS Fundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Manero G, McCloskey J, Griffiths EA, Yee KWL, Zeidan AM, Al-Kali A, Deeg HJ, Patel PA, Sabloff M, Keating MM, Zhu N, Gabrail NY, Fazal S, Maly J, Odenike O, Kantarjian H, DeZern AE, O'Connell CL, Roboz GJ, Busque L, Buckstein R, Amin H, Randhawa J, Leber B, Shastri A, Dao KH, Oganesian A, Hao Y, Keer HN, Azab M, Savona MR. Oral decitabine-cedazuridine versus intravenous decitabine for myelodysplastic syndromes and chronic myelomonocytic leukaemia (ASCERTAIN): a registrational, randomised, crossover, pharmacokinetics, phase 3 study. Lancet Haematol. 2024 Jan;11(1):e15-e26. doi: 10.1016/S2352-3026(23)00338-1. PMID 38135371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 227 participants took part in the study from 15 February 2018 to 25 May 2023. 138 participants with a diagnosis of myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) took part from the United States and Canada. 89 participants with a diagnosis of acute myeloid leukemia (AML) took part from Austria, Canada, Czech Republic, France, Germany, Hungary, Italy, Spain, and United Kingdom.
Pre-assignment Details: A total of 138 participants with a diagnosis of MDS or CMML were enrolled and randomized in a 1:1 ratio to receive ASTX727 or decitabine in a crossover manner. A total of 89 participants with a diagnosis of AML were enrolled and randomized in a 1:1 ratio to receive ASTX727 or decitabine in a crossover manner.
Period: Overall Study
Arm/Group | MDS or CMML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | MDS or CMML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727 | AML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | AML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727
Started | 69 | 69 | 44 | 45
Safety Analysis Set (The Safety Analysis Set included all participants who received any amount of study treatment.) | 66 | 67 | 43 | 44
Completed | 0 | 0 | 0 | 0
Not Completed | 69 | 69 | 44 | 45
Not completed — Death | 33 | 25 | 34 | 34
Not completed — Complete Consent Withdrawal | 4 | 4 | 1 | 8
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Rollover to ASTX727-06 | 10 | 18 | 4 | 2
Not completed — Study Centre Terminated by Sponsor | 21 | 22 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received any amount of study treatment.
Groups:
- MDS or CMML: ASTX727 or IV Decitabine: Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2 or the converse. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
- AML: ASTX727 or IV Decitabine: Participants with AML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2 or the converse. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
- Total: Total of all reporting groups
Arm/Group | MDS or CMML: ASTX727 or IV Decitabine | AML: ASTX727 or IV Decitabine | Total
Number analyzed (Participants) | 133 | 87 | 220
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 36 | 3 | 39
  65 to 84 years | 93 | 75 | 168
  ≥85 years | 4 | 9 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 34 | 80
  Male | 87 | 53 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 125 | 0 | 125
  Unknown or Not Reported | 2 | 87 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 121 | 0 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 87 | 92

OUTCOME MEASURES:

1. Primary Outcome: Total 5-day Area Under the Curve From 0 to 24 Hours (AUC0-24) After Treatment With ASTX727 And IV Decitabine
Description: Total 5-day ASTX727 AUC0-24 exposures were calculated using PK data from 3 days of serial PK sampling, Day 1 AUC0-24 (first ASTX727 dose) was added to (Day 2 AUC0-24+ Day 5 AUC0-24) × 2. Decitabine 5-day AUC0-24 exposures after IV decitabine were calculated as follows: (Day 1 AUC0-24+ Day 5 AUC0-24) / 2 was multiplied by 5. If AUC0-24 on Day 2 (for ASTX727) or Day 1 (IV decitabine) was not available, it was replaced by AUC0-24 on Day 5; the converse was also true.
Time Frame: ASTX727: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose on Days 1 to 5 of Cycle 1 and 2; Decitabine: Pre-dose, 0.25, 0.5, 1, 1.08, 1.5, 2, 3, 4, 6, 8 hours post-dose on Days 1 to 5 of Cycle 1 and 2 (each cycle= 28 days)
Population: Primary Endpoint Pharmacokinetics (PK) Analysis Set included participants who received full dose of ASTX727 within 3 hours of the intended dosing time, and no vomiting within 6 hours of dosing, and had at least 2 days of evaluable decitabine (AUC0-24) measurements in the ASTX727 cycle, i.e, Day 1 and either Day 2 or Day 5 and received the full IV decitabine dose as a 1-hour infusion.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Groups:
- MDS or CMML: IV Decitabine: Participants with MDS or CMML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle=28 days).
- MDS or CMML: ASTX727: Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle = 28 days). From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
- AML: IV Decitabine: Participants with AML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle=28 days).
- AML: ASTX727: Participants with AML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle = 28 days). From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 123 | 123 | 69 | 69
hours*nanograms per milliliter (h*ng/mL) | 864.34 (40.0) | 855.96 (50.6) | 910.1 (52.4) | 900.5 (52.0)
Statistical Analysis 1: Comparison: MDS or CMML: IV Decitabine vs MDS or CMML: ASTX727; MDS or CMML: IV Decitabine Versus MDS or CMML: ASTX727; Test type: Equivalence — ASTX727 and IV decitabine were to be considered equivalent if the 2-sided 90% confidence interval (CI) of the 5-day AUC0-24 ratio of Least Square Mean (LSM) for oral/IV was contained entirely within the range of 0.80 - 1.25; Ratio of Geometric LSM = 98.93, 90% CI 2-sided [92.66 to 105.6] — Analysis was based on ANOVA model with treatment, cycle, and sequence as fixed effects, and participant nested in sequence as a random effect (ratio is Oral/IV)
Statistical Analysis 2: Comparison: AML: IV Decitabine vs AML: ASTX727; AML: IV Decitabine Versus AML: ASTX727; Test type: Equivalence — ASTX727 and IV decitabine were to be considered equivalent if the 2-sided 90% CI of the 5-day AUC0-24 ratio of LSM for oral/IV was contained entirely within the range of 0.80 - 1.25; Ratio of Geometric LSM = 99.64, 90% CI 2-sided [91.23 to 108.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: MDS/CMML: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participants administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs were defined as events that first occurred or worsened on or after the date of the first dose of study treatment until 30 days after the last dose of study treatment or until the start of a post-treatment alternative anti-cancer treatment, whichever occurred first.
Time Frame: From randomization up to 30 days after last dose of study treatment (up to approximately 2.7 years)
Population: The Safety Analysis Set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727
Number analyzed (Participants) | 132 | 130
Participants | 127 | 130

3. Secondary Outcome: AML: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: as for outcome 2
Time Frame: From randomization up to 30 days after last dose of study treatment (up to approximately 2.4 years)
Population: The Safety Analysis Set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 78 | 80
Participants | 71 | 80

4. Secondary Outcome: MDS/CMML: Number of Participants With Grade 3 or Higher TEAEs
Description: TEAEs were defined as events that first occurred or worsened on or after the date of the first dose of study treatment until 30 days after the last dose of study treatment or until the start of a post-treatment alternative anti-cancer treatment, whichever occurred first. Severity of AEs were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal.
Time Frame: From randomization up to 30 days after last dose of study treatment (up to approximately 2.7 years)
Population: The Safety Analysis Set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- MDS or CMML: IV Decitabine: Participants with MDS or CMML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle = 28 days).
- MDS or CMML: ASTX727: Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days). From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727
Number analyzed (Participants) | 132 | 130
Participants | 89 | 121

5. Secondary Outcome: AML: Number of Participants With Grade 3 or Higher TEAEs
Description: TEAEs were defined as events that first occurred or worsened on or after the date of the first dose of study treatment until 30 days after the last dose of study treatment or until the start of a post-treatment alternative anti-cancer treatment, whichever occurred first. Severity of AEs were graded using CTCAE version 4.03. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Fatal.
Time Frame: From randomization up to 30 days after last dose of study treatment (up to approximately 2.4 years)
Population: The Safety Analysis Set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- AML: IV Decitabine: Participants with AML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle = 28 days).
- AML: ASTX727: Participants with AML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days). From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
Arm/Group | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 78 | 80
Participants | 43 | 73

6. Secondary Outcome: Maximum Percentage of Long Interspersed Nucleotide Elements (LINE)-1 Demethylation
Description: Summarized data for Cycle 1 and Cycle 2 was reported.
Time Frame: Pre-dose on Day 1 of Cycles 1 and 2 (as Baseline), and Days 8, 15 and 22 of Cycles 1 and 2 (each cycle= 28 days)
Population: Pharmacodynamic (PD) LINE-1 Analysis Set included participants who received any amount of study treatment and have LINE-1 methylation data at baseline (Day 1) of Cycle 1 or 2 and on either Day 8 or Day 15 of the respective cycle. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure. 'Number analyzed' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of demethylation
Groups:
- MDS or CMML: IV Decitabine: Participants with MDS or CMML received decitabine 20 mg/m^2 IV injection, once daily, on Days 1 to 5 in cycle 1 or 2 (each cycle = 28 days).
- MDS or CMML: ASTX727: Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, given by mouth, once daily, on Days 1 to 5 in cycle 1 or 2 (each cycle = 28 days). From cycle 3, participants received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
- AML: IV Decitabine: Participants with AML received decitabine 20 mg/m^2 IV injection, once daily, on Days 1 to 5 in cycle 1 or 2 (each cycle = 28 days).
- AML: ASTX727: Participants with AML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, given by mouth, once daily, on Days 1 to 5 in cycle 1 or 2 (each cycle = 28 days). From cycle 3, participants received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 63 | 63 | 39 | 34
percentage of demethylation
  Cycle 1: number analyzed (Participants) | 62 | 62 | 39 | 33
  Cycle 1 | 14.019 [12.528 to 15.510] | 13.289 [11.798 to 14.780] | 8.243 [6.340 to 10.147] | 9.357 [7.288 to 11.426]
  Cycle 2: number analyzed (Participants) | 63 | 63 | 29 | 34
  Cycle 2 | 11.968 [10.503 to 13.434] | 11.151 [9.685 to 12.616] | 8.153 [6.226 to 10.079] | 8.037 [6.258 to 9.816]

7. Secondary Outcome: Total 5-day Area Under the Curve From 0 to Infinity (AUC0-inf) After Treatment With ASTX727 And IV Decitabine
Description: Total 5-day ASTX727 AUC0-inf exposures were calculated using PK data from 3 days of serial PK sampling, Day 1 AUC0-inf (first ASTX727 dose) was added to (Day 2 AUC0-inf+ Day 5 AUC0-inf) × 2. Decitabine 5-day AUC0-inf exposures after IV decitabine were calculated as follows: (Day 1 AUC0-inf+ Day 5 AUC0-inf) / 2 was multiplied by 5. If AUC0-inf on Day 2 (for ASTX727) or Day 1 (IV decitabine) was not available, it was replaced by AUC0-inf on Day 5; the converse was also true.
Time Frame: as for outcome 1
Population: Overall PK Analysis Set included participants who may not have been included in the Primary Endpoint PK Analysis Set and who received any amount of study treatment, complied with the protocol sufficiently to ensure PK samples were collected as intended and provided sufficient samples to measure available plasma concentrations for decitabine. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 123 | 123 | 69 | 69
h*ng/mL | 866.15 (39.9) | 849.63 (50.4) | 912.3 (52.3) | 902.1 (51.8)
Statistical Analysis 1: Comparison: MDS or CMML: IV Decitabine vs MDS or CMML: ASTX727; MDS or CMML: IV Decitabine Versus MDS or CMML: ASTX727; Test type: Equivalence — ASTX727 and IV decitabine were to be considered equivalent if the 2-sided 90% CI of the 5-day AUC0-inf ratio of LSM for oral/IV was contained entirely within the range of 0.80 - 1.25; Ratio of Geometric LSM = 98.00, 90% CI 2-sided [91.80 to 104.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AML: IV Decitabine vs AML: ASTX727; AML: IV Decitabine Versus AML: ASTX727; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio of Geometric LSM = 99.61, 90% CI 2-sided [91.20 to 108.8] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Total 5-day Area Under the Curve From 0 to Last Quantifiable Concentration (AUC0-last) After Treatment With ASTX727 And IV Decitabine
Description: Total 5-day ASTX727 AUC0-last exposures were calculated using PK data from 3 days of serial PK sampling, Day 1 AUC0-last (first ASTX727 dose) was added to (Day 2 AUC0-last + Day 5 AUC0-last) × 2. Decitabine 5-day AUC0-last exposures after IV decitabine were calculated as follows: (Day 1 AUC0-last + Day 5 AUC0-last) / 2 was multiplied by 5. If AUC0-last on Day 2 (for ASTX727) or Day 1 (IV decitabine) was not available, it was replaced by AUC0-last on Day 5; the converse was also true.
Time Frame: as for outcome 1
Population: Overall PK Analysis Set included participants who may not have been included in the Primary Endpoint PK Analysis Set and received any amount of study treatment, complied with the protocol sufficiently to ensure PK samples were collected as intended and provided sufficient samples to measure available plasma concentrations for decitabine. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 124 | 124 | 70 | 70
h*ng/mL | 853.02 (40.7) | 837.38 (50.7) | 902.7 (53.0) | 881.8 (52.5)
Statistical Analysis 1: Comparison: MDS or CMML: IV Decitabine vs MDS or CMML: ASTX727; MDS or CMML: IV Decitabine Versus MDS or CMML: ASTX727; Test type: Equivalence — ASTX727 and IV decitabine were to be considered equivalent if the 2-sided 90% CI of the 5-day AUC0-last ratio of LSM for oral/IV was contained entirely within the range of 0.80 - 1.25; Ratio of Geometric LSM = 98.11, 90% CI 2-sided [91.88 to 104.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AML: IV Decitabine vs AML: ASTX727; AML: IV Decitabine Versus AML: ASTX727; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; Ratio of Geometric LSM = 98.11, 90% CI 2-sided [89.75 to 107.2] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Total 5-day Area Under the Curve From 0 to 8 Hours (AUC0-8) After Treatment With ASTX727 And IV Decitabine
Description: Total 5-day ASTX727 AUC0-8 exposures were calculated using PK data from 3 days of serial PK sampling, Day 1 AUC0-8 (first ASTX727 dose) was added to (Day 2 AUC0-8 + Day 5 AUC0-8) × 2. Decitabine 5-day AUC0-8 exposures after IV decitabine were calculated as follows: (Day 1 AUC0-8 + Day 5 AUC0-8) / 2 was multiplied by 5. If AUC0-8 on Day 2 (for ASTX727) or Day 1 (IV decitabine) was not available, it was replaced by AUC0-8 on Day 5; the converse was also true.
Time Frame: ASTX727: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post-dose on Days 1 to 5 of Cycle 1 and 2; Decitabine: Pre-dose, 0.25, 0.5, 1, 1.08, 1.5, 2, 3, 4, 6, 8 hours post-dose on Days 1 to 5 of Cycle 1 and 2 (each cycle= 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 124 | 124 | 70 | 70
h*ng/mL | 856.63 (40.6) | 839.37 (50.4) | 910.1 (52.0) | 883.8 (52.1)
Statistical Analysis 1: Comparison: MDS or CMML: IV Decitabine vs MDS or CMML: ASTX727; MDS or CMML: IV Decitabine Versus MDS or CMML: ASTX727; Test type: Equivalence — ASTX727 and IV decitabine were to be considered equivalent if the 2-sided 90% CI of the 5-day AUC0-8 ratio of LSM for oral/IV was contained entirely within the range of 0.80 - 1.25; Ratio of Geometric LSM = 97.93, 90% CI 2-sided [91.74 to 104.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AML: IV Decitabine vs AML: ASTX727; AML: IV Decitabine Versus AML: ASTX727; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Ratio of Geometric LSM = 97.55, 90% CI 2-sided [89.32 to 106.5] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Area Under the Curve From 0 to Infinity (AUC0-inf) After Treatment With ASTX727 And IV Decitabine
Description: AUC0-inf was calculated using the formula AUClast + (Clast / λZ), where Clast is the last quantifiable concentration and λZ is the elimination rate constant. AUC0-inf will be calculated using the linear up-log down method. Summarized data has been reported for cycle 1 and 2.
Time Frame: ASTX727: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose on Days 1, 2 and 5 of Cycle 1 and 2; Decitabine: Pre-dose, 0.25, 0.5, 1, 1.08, 1.5, 2, 3, 4, 6, 8 hours post-dose on Days 1 and 5 of Cycle 1 and 2 (each cycle= 28 days)
Population: Overall PK Analysis Set included participants not included in Primary Endpoint PK Analysis Set, received any amount of study treatment, complied with protocol sufficiently to ensure PK samples were collected, provided sufficient samples to measure available plasma concentrations for decitabine. Overall number of participants analyzed:Number of participants evaluable for this outcome measure. Number analyzed:Number of participants evaluable for this outcome measure at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per millilitres(ng*h/mL)
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 119 | 127 | 70 | 78
nanograms*hours per millilitres(ng*h/mL)
  Day 1 | 174 (40.8) | 102 (54.8) | 175 (54.9) | 118 (54.4)
  Day 2: number analyzed (Participants) | 0 | 126 | 0 | 74
  Day 2 |  | 186 (55.3) |  | 193 (59.6)
  Day 5: number analyzed (Participants) | 119 | 123 | 70 | 75
  Day 5 | 170 (41.7) | 178 (52.7) | 181 (58.1) | 187 (57.1)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Decitabine, Cedazuridine, and Cedazuridine-epimer
Description: Summarized data of Cmax on Day 1, 2 and 5 respectively for Cycle 1 and 2 has been reported for ASTX727. Similarly, summarized data of Cmax on Day 1 and 5 respectively for Cycle 1 and 2 has been reported for IV Decitabine.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 122 | 128 | 72 | 79
nanogram per milliliter (ng/mL)
  Decitabine: Day 1: number analyzed (Participants) | 122 | 128 | 72 | 78
  Decitabine: Day 1 | 184 (48.1) | 83.1 (66.1) | 187 (64.7) | 85.9 (56.6)
  Decitabine: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 76
  Decitabine: Day 2 |  | 145 (54.7) |  | 139 (58.5)
  Decitabine: Day 5: number analyzed (Participants) | 122 | 124 | 70 | 76
  Decitabine: Day 5 | 180 (49.2) | 140 (62.8) | 192 (62.4) | 139 (62.7)
  Cedazuridine: Day 1: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine: Day 1 |  | 321 (53.8) |  | 313 (47.7)
  Cedazuridine: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine: Day 2 |  | 349 (49.1) |  | 343 (43.4)
  Cedazuridine: Day 5: number analyzed (Participants) | 0 | 126 | 0 | 77
  Cedazuridine: Day 5 |  | 371 (51.8) |  | 350 (42.7)
  Cedazuridine-epimer: Day 1: number analyzed (Participants) | 0 | 128 | 0 | 79
  Cedazuridine-epimer: Day 1 |  | 150 (65.7) |  | 182 (60.0)
  Cedazuridine-epimer: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine-epimer: Day 2 |  | 155 (64.6) |  | 204 (59.2)
  Cedazuridine-epimer: Day 5: number analyzed (Participants) | 0 | 126 | 0 | 77
  Cedazuridine-epimer: Day 5 |  | 169 (65.9) |  | 191 (58.4)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Decitabine, Cedazuridine, and Cedazuridine-epimer
Description: Summarized data of Tmax on Day 1, 2 and 5 respectively for Cycle 1 and 2 has been reported for ASTX727. Similarly, summarized data of Tmax on Day 1 and 5 respectively for Cycle 1 and 2 has been reported for IV Decitabine.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 122 | 128 | 72 | 79
hours
  Decitabine: Day 1: number analyzed (Participants) | 122 | 128 | 72 | 78
  Decitabine: Day 1 | 0.98 [0.23 to 1.27] | 1.00 [0.48 to 3.00] | 0.98 [0.25 to 2.00] | 1.00 [0.25 to 2.02]
  Decitabine: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 76
  Decitabine: Day 2 |  | 1.00 [0.47 to 2.00] |  | 1.00 [0.25 to 3.00]
  Decitabine: Day 5: number analyzed (Participants) | 122 | 124 | 70 | 76
  Decitabine: Day 5 | 0.97 [0.25 to 1.62] | 1.00 [0.25 to 3.00] | 0.98 [0.00 to 1.17] | 1.00 [0.47 to 3.00]
  Cedazuridine: Day 1: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine: Day 1 |  | 3.00 [1.50 to 7.97] |  | 3.98 [1.47 to 8.00]
  Cedazuridine: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine: Day 2 |  | 3.01 [0.52 to 7.88] |  | 4.00 [1.00 to 7.88]
  Cedazuridine: Day 5: number analyzed (Participants) | 0 | 126 | 0 | 77
  Cedazuridine: Day 5 |  | 3.00 [1.50 to 6.12] |  | 3.98 [1.00 to 8.00]
  Cedazuridine-epimer: Day 1: number analyzed (Participants) | 0 | 128 | 0 | 79
  Cedazuridine-epimer: Day 1 |  | 3.08 [1.50 to 7.97] |  | 4.00 [1.50 to 8.03]
  Cedazuridine-epimer: Day 2: number analyzed (Participants) | 0 | 128 | 0 | 78
  Cedazuridine-epimer: Day 2 |  | 3.03 [0.52 to 7.88] |  | 4.00 [1.50 to 7.88]
  Cedazuridine-epimer: Day 5: number analyzed (Participants) | 0 | 126 | 0 | 77
  Cedazuridine-epimer: Day 5 |  | 3.08 [1.00 to 8.05] |  | 4.00 [1.53 to 8.00]

13. Secondary Outcome: Apparent Oral Clearance (CL/F) of Oral Decitabine and Cedazuridine
Description: Oral CL/F for oral decitabine was measured only on Day 1 and oral CL/F for oral cedazuridine was measured on Days 1, 2 and 5. Summarized data of Oral CL/F for oral decitabine on Day 1 for Cycle 1 and 2 has been reported for ASTX727. Similarly, summarized data of oral CL/F for oral cedazuridine on Day 1,2 and 5 respectively for Cycle 1 and 2 has been reported for ASTX727.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose on Days 1, 2 and 5 of Cycle 1 and 2 (each cycle= 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | MDS or CMML: ASTX727 | AML: ASTX727
Number analyzed (Participants) | 127 | 78
Litres per hour (L/h)
  Decitabine: Day 1 | 342 (54.8) | 297 (54.4)
  Cedazuridine: Day 1: number analyzed (Participants) | 109 | 52
  Cedazuridine: Day 1 | 30.6 (46.4) | 28.6 (55.5)
  Cedazuridine: Day 2: number analyzed (Participants) | 121 | 74
  Cedazuridine: Day 2 | 25.6 (159) | 27.4 (45.4)
  Cedazuridine: Day 5: number analyzed (Participants) | 2 | 1
  Cedazuridine: Day 5 | 16.8 (15.9) | 86.8 (NA) — Geometric Coefficient of Variation could not be calculated as data for only one participant was available for analysis.

14. Secondary Outcome: Apparent Elimination Half Life (t1/2) of Decitabine, Cedazuridine, and Cedazuridine-epimer
Description: Summarized data of t1/2 on Day 1, 2 and 5 respectively for Cycle 1 and 2 has been reported for ASTX727. Similarly, summarized data of t1/2 on Day 1 and 5 respectively for Cycle 1 and 2 has been reported for IV Decitabine.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | AML: IV Decitabine | AML: ASTX727
Number analyzed (Participants) | 119 | 127 | 70 | 78
hours
  Decitabine: Day 1 | 0.967 (46.8) | 1.18 (22.8) | 1.16 (56.7) | 1.07 (31.6)
  Decitabine: Day 2: number analyzed (Participants) | 0 | 126 | 0 | 74
  Decitabine: Day 2 |  | 1.38 (24.7) |  | 1.36 (35.0)
  Decitabine: Day 5: number analyzed (Participants) | 119 | 123 | 70 | 75
  Decitabine: Day 5 | 1.14 (44.9) | 1.47 (26.9) | 1.18 (49.0) | 1.45 (34.0)
  Cedazuridine: Day 1: number analyzed (Participants) | 0 | 109 | 0 | 52
  Cedazuridine: Day 1 |  | 6.33 (18.1) |  | 6.68 (18.5)
  Cedazuridine: Day 2: number analyzed (Participants) | 0 | 115 | 0 | 56
  Cedazuridine: Day 2 |  | 6.70 (18.9) |  | 7.05 (17.6)
  Cedazuridine: Day 5: number analyzed (Participants) | 0 | 2 | 0 | 1
  Cedazuridine: Day 5 |  | 2.59 (5.43) |  | 2.41 (NA) — Geometric Coefficient of Variation could not be calculated as data for only one participant was available for analysis.
  Cedazuridine-epimer: Day 1: number analyzed (Participants) | 0 | 107 | 0 | 49
  Cedazuridine-epimer: Day 1 |  | 5.50 (21.8) |  | 6.22 (17.4)
  Cedazuridine-epimer: Day 2: number analyzed (Participants) | 0 | 105 | 0 | 45
  Cedazuridine-epimer: Day 2 |  | 5.90 (23.2) |  | 6.15 (22.8)
  Cedazuridine-epimer: Day 5: number analyzed (Participants) | 0 | 9 | 0 | 1
  Cedazuridine-epimer: Day 5 |  | 2.58 (5.16) |  | 2.57 (NA) — Geometric Coefficient of Variation could not be calculated as data for only one participant was available for analysis.

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Oral Decitabine and Cedazuridine
Description: Summarized data of Vz/F on Day 1, 2 and 5 respectively for Cycle 1 and 2 has been reported for ASTX727.
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | MDS or CMML: ASTX727 | AML: ASTX727
Number analyzed (Participants) | 127 | 78
Litres
  Decitabine: Day 1 | 585 (55.0) | 434 (60.4)
  Decitabine: Day 2: number analyzed (Participants) | 126 | 74
  Decitabine: Day 2 | 369 (59.0) | 337 (67.6)
  Decitabine: Day 5: number analyzed (Participants) | 123 | 75
  Decitabine: Day 5 | 417 (54.3) | 373 (68.9)
  Cedazuridine: Day 1: number analyzed (Participants) | 109 | 52
  Cedazuridine: Day 1 | 280 (50.9) | 272 (59.9)
  Cedazuridine: Day 2: number analyzed (Participants) | 118 | 56
  Cedazuridine: Day 2 | 296 (51.3) | 278 (49.8)
  Cedazuridine: Day 5: number analyzed (Participants) | 2 | 1
  Cedazuridine: Day 5 | 62.8 (10.4) | 302 (NA) — Geometric Coefficient of Variation could not be calculated as data for only one participant was available for analysis.

16. Secondary Outcome: MDS/CMML: Percentage of Participants With Complete Response (CR), Marrow CR (mCR), Partial Response (PR), Hematologic Improvement (HI) Based on International Working Group (IWG) 2006 Myelodysplastic Syndromes (MDS) Response Criteria
Description: CR: normal peripheral, persistent granulocyte count ≥1.0x10^9/liter(L), platelet ≥100x10^9/L, Hemoglobin (Hgb) ≥11g/dL, normal bone marrow with persistent marrow blasts ≤5%. mCR: reduction of bone marrow blasts to≤5%, decrease by 50% or more with/without normalization of peripheral counts.PR: normal peripheral counts, granulocyte count ≥1.0x10^9/L, platelet count ≥100x10^9/L, Hgb ≥11 g/dL, normal bone marrow, marrow blasts >5%, reduced by 50% or more for at least 4 weeks. HI: HI-E: Hb increase ≥1.5 g/dL in absence of RBC transfusions. HI-P: Absolute increase of platelet count from <20 to >20X10^9/L by at least 100%,if more than 20x10^9/L, by absolute increase of at least 30x10^9/L in absence of platelet transfusions. HI-N: granulocyte increase ≥100%, by an absolute increase ≥0.5x10^9/L for at least 8 weeks. Percentage of participants with CR, mCR, PR, and HI based on IWG 2003 MDS response criteria are reported. Response has been reported based on participants with MDS or CMML.
Time Frame: Up to approximately 2.7 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MDS: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727: Participants with MDS received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
- MDS: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727: Participants with MDS received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days) followed by ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
- CMML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727: Participants with CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days), followed by IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
- CMML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727: Participants with CMML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycle 1 (each cycle = 28 days) followed by ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycle 2. A washout period of 23 days was maintained between the 2 cycles. From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, treatment discontinuation for other reasons, or withdrawal from the study.
Arm/Group | MDS: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | MDS: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727 | CMML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | CMML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727
Number analyzed (Participants) | 61 | 56 | 5 | 11
percentage of participants
  Complete Response (CR) | 26.2 [15.8 to 39.1] | 19.6 [10.2 to 32.4] | 0 [0 to 0] | 18.2 [2.3 to 51.8]
  Marrow Complete Response (mCR) | 29.5 [18.5 to 42.6] | 30.4 [18.8 to 44.1] | 40.0 [5.3 to 85.3] | 54.5 [23.4 to 83.3]
  Partial Response (PR) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  HI: Erythroid Response (HI-E) | 0 [0 to 0] | 1.8 [0.0 to 9.6] | 20.0 [0.5 to 71.6] | 0 [0 to 0]
  HI: Platelet Response (HI-P) | 3.3 [0.4 to 11.3] | 8.9 [3.0 to 19.6] | 0 [0 to 0] | 0 [0 to 0]
  HI: Neutrophil Response (HI-N) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 9.1 [0.2 to 41.3]

17. Secondary Outcome: AML: Percentage of Participants With CR, CR With Incomplete Blood Count Recovery (CRi), CR With Incomplete Platelet Recovery (CRp), and CR Plus CRp Based on IWG 2003 AML Response Criteria
Description: CR was defined as absolute neutrophil content (ANC) ≥1000/ microliter (μL), platelets ≥100,000/μL, independence from red blood cell (RBC) and platelet transfusions over the past week, no leukemic blasts and <5% leukemic blasts. CRp was defined as CR criteria except platelets <100,000/μL.and platelet transfusion over the past week. CRi was defined as CR criteria except ANC <1000/μL or platelets <100,000/μL. Percentage of participants with CR, CRi, CRp, and CR Plus CRp based on IWG 2003 AML response criteria are reported.
Time Frame: Up to approximately 2.4 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | AML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727
Number analyzed (Participants) | 43 | 44
percentage of participants
  Complete Response (CR) | 14.0 [5.3 to 27.9] | 29.5 [16.8 to 45.2]
  CR with Incomplete Platelet Recovery (CRp) | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.0]
  CR with Incomplete Blood Count Recovery (CRi) | 11.6 [3.9 to 25.1] | 0 [0.0 to 8.0]
  CR Plus CRp | 18.6 [8.4 to 33.4] | 29.5 [16.8 to 45.2]

18. Secondary Outcome: AML: Percentage of Participants With CR With Partial Hematologic Recovery (CRh) Based on IWG 2003 AML Response Criteria
Description: CRh was defined as <5% of blasts in the bone marrow, no evidence of disease, and partial recovery of peripheral blood counts (platelets >50,000/μL and ANC >500/μL), independence from RBC and platelet transfusions within 7 days of bone marrow evaluation, and peripheral blast ≤1%. Percentage of participants with CRh based on IWG 2003 AML response criteria are reported.
Time Frame: Day 1 of Cycle 3 up to approximately 2.4 years (each cycle= 28 days)
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AML: Sequence A: First ASTX727, Then IV Decitabine, Then ASTX727 | AML: Sequence B: First IV Decitabine, Then ASTX727, Then ASTX727
Number analyzed (Participants) | 43 | 44
percentage of participants | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.0]

19. Secondary Outcome: AML: Time to First Response, Best Response and Complete Response Based on IWG 2003 AML Response Criteria
Description: Time to first response was defined as time in months from the date of first treatment to the first date when any response is achieved. Time to best response was defined in months from the date of first treatment to the first date when a subject's best response, in the order of CR, CRi (or CRp or CRh), or PR, was achieved. Time to CR was defined in months from the date of first treatment to the first date when CR is achieved. CR:ANC ≥1000/ microliter (μL),platelets ≥100,000/μL,independence from RBC and platelet transfusions over the past week, no leukemic blasts, and <5% leukemic blasts.CRp: CR criteria except ANC ≥1000/μL, platelets < 100,000/μL.and platelet transfusion over the past week. CRi:CR criteria except ANC <1000/μL or platelets <100,000/μL.CRh: <5% of blasts in the bone marrow,platelets >50,000/μL and ANC >500/μL, independence from RBC and platelet transfusions within 7 days and peripheral blast ≤1%. PR: CR criteria except decrease of ≥50% in leukemic blasts.
Time Frame: Up to approximately 2.4 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 87
months
  Time to First Response | 2.91 [1.9 to 6.5]
  Time to Best Response | 3.45 [1.9 to 7.5]
  Time to Complete Response | 3.02 [1.9 to 7.5]

20. Secondary Outcome: AML: Duration of Complete Response and Combined CR and CRh Based on IWG 2003 AML Response Criteria
Description: Duration of CR was defined as the time interval from the first CR to time of relapse. Duration of combined CR and CRh was defined as the time interval from the first CR or CRh to time of relapse. Duration of CR and combined CR and CRh was presented using a Kaplan-Meier estimate.
Time Frame: Up to approximately 2.4 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 87
months
  Duration of Complete Response | 6.9 [3.4 to 11.5]
  Duration of Combined CR and CRh | 9.0 [3.4 to 11.5]

21. Secondary Outcome: MDS/CMML: Percentage of Participants With Red Blood Cell (RBC) and Platelet Transfusion Independence (TI)
Description: Transfusion independence was defined as no transfusion for 56 consecutive days or more (84 and 112 days) after the first dose of study treatment while maintaining hemoglobin ≥8 grams/deciliter (g/dL) (RBC TI) or maintaining platelets ≥20×109/L (platelet TI).
Time Frame: Up to approximately 2.7 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure. 'Number analyzed' signifies those subjects who were evaluable for this outcome measure in specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MDS or CMML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 54
percentage of participants
  RBC TI: ≥56 Days | 51.9 [37.8 to 65.7]
  RBC TI: ≥84 Days | 40.7 [27.6 to 55.0]
  RBC TI: ≥112 Days | 33.3 [21.1 to 47.5]
  Platelet TI: ≥56 Days: number analyzed (Participants) | 12
  Platelet TI: ≥56 Days | 50.0 [21.1 to 78.9]
  Platelet TI: ≥84 Days: number analyzed (Participants) | 12
  Platelet TI: ≥84 Days | 33.3 [9.9 to 65.1]
  Platelet TI: ≥112 Days: number analyzed (Participants) | 12
  Platelet TI: ≥112 Days | 33.3 [9.9 to 65.1]

22. Secondary Outcome: AML: Percentage of Participants With Red Blood Cell (RBC) and Platelet Transfusion Independence (TI)
Description: Transfusion independence was defined as no transfusion for 56 consecutive days or more (112 days) after the first dose of study treatment while maintaining hemoglobin ≥8 grams/deciliter (g/dL) (RBC TI) or maintaining platelets ≥20×109/L (platelet TI).
Time Frame: Up to approximately 2.4 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure. 'Number analyzed' signifies those subjects who were evaluable for this outcome measure at specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 37
percentage of participants
  RBC TI ≥56 Days | 37.8 [22.5 to 55.2]
  RBC TI ≥112 Days | 24.3 [11.8 to 41.2]
  Platelet TI ≥56 Days: number analyzed (Participants) | 14
  Platelet TI ≥56 Days | 35.7 [12.8 to 64.9]
  Platelet TI ≥112 Days: number analyzed (Participants) | 14
  Platelet TI ≥112 Days | 28.6 [8.4 to 58.1]

23. Secondary Outcome: MDS/CMML: Leukemia-free Survival (LFS)
Description: LFS was defined as time from the date of randomization to the date when bone marrow or peripheral blood blasts reach ≥20%, or death from any cause. Participants who hadn't reached AML at the time of the analysis were censored at the date of the last follow-up. Leukemia-free survival was presented using a Kaplan-Meier estimate.
Time Frame: From randomization up to approximately 2.7 years
Population: Efficacy Analysis Set included all participants who received any amount of study treatment. 'Overall number of participants analyzed' signifies those who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MDS or CMML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 62
days | 889.0 [674.0 to NA] — The upper limit of the 95% Confidence Interval (CI) was not reached at time of data cut-off due to insufficient number of participants with an event.

24. Secondary Outcome: MDS/CMML: Overall Survival (OS)
Description: OS was defined as time from the date of randomization to the date of death from any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. Overall survival was presented using a Kaplan-Meier estimate.
Time Frame: From randomization up to approximately 2.7 years
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MDS or CMML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 58
days | 966.0 [809.0 to NA] — The upper limit of the 95% CI was not reached at time of data cut-off due to insufficient number of participants with an event.

25. Secondary Outcome: AML: Overall Survival (OS)
Description: as for outcome 24
Time Frame: From randomization up to approximately 2.4 years
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 67
months | 8.9 [5.9 to 13.1]

26. Secondary Outcome: AML: Survival Rates at 6 Months, 1 Year, and 2 Years
Description: One-year survival rate was defined as the survival rate at the end of the first year from the date of randomization. The survival rates at 6 months and at 2 years were calculated similarly.
Time Frame: At Month 6, Year 1 and 2
Population: Efficacy Analysis Set included all participants who received any amount of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 87
percentage of participants
  Month 6 | 61 [50 to 71]
  Year 1 | 44 [33 to 54]
  Year 2 | 16 [8 to 26]

27. Secondary Outcome: AML: Event-free Survival (EFS)
Description: EFS was defined as time from the date of randomization to the date of treatment failure [disease progression/relapse (due to confirmed reappearance of leukemic blasts in peripheral blood or ≥5% leukemic blasts in bone marrow (including relapse), discontinue treatment due to disease progression or treatment-related AE, or alternative anti-leukemia therapy except for HCT] or death from any cause, whichever occurs first. Participants without documented treatment failure at the time of the analysis were censored at the date of the last follow-up. Event-free survival was presented using a Kaplan-Meier estimate.
Time Frame: From randomization up to approximately 2.4 years
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 82
months | 5.9 [3.8 to 8.5]

28. Secondary Outcome: AML: Progression-free Survival (PFS)
Description: PFS was defined as time from the date of randomization to the date disease progression due to confirmed reappearance of leukemic blasts in peripheral blood or ≥5% leukemic blasts in bone marrow (including relapse) or death from any cause, whichever occurs first. Participants without documented disease progression/relapse or death at the time of the analysis were censored at the date of the last follow-up. Progression-free survival was presented using a Kaplan-Meier estimate.
Time Frame: From randomization up to approximately 2.4 years
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AML: ASTX727 or IV Decitabine
Number analyzed (Participants) | 78
months | 6.1 [4.0 to 8.7]

ADVERSE EVENTS:
Time Frame: MDS or CMML: From randomization up to 2.7 years; AML: From randomization up to 2.4 years
Description: All-cause mortality: Randomized Analysis Set included all randomized participants. Serious adverse events and non-serious adverse events: Safety Analysis Set included all participants who received any amount of study treatment.
Groups:
- MDS or CMML: ASTX727: Participants with MDS or CMML received ASTX727 tablet, containing the fixed-dose combination of 35 mg decitabine and 100 mg cedazuridine, orally, once daily, on Days 1 to 5 in cycles 1 or 2 (each cycle = 28 days). From cycle 3, all participants enrolled in cycles 1 and 2 received ASTX727 tablet, once daily, on Days 1 to 5 of each 28-day cycle until disease progression, unacceptable toxicity, participant discontinued treatment, or was withdrawn from the study.
- MDS or CMML: Not Treated: Participants with MDS or CMML were enrolled in the study but did not receive any study treatment.
- AML: IV Decitabine: Participants with MDS or CMML received IV infusion of decitabine 20 mg/m^2, once daily, on Days 1 to 5 in cycles 1 or 2.
- AML: Not Treated: Participants with AML were enrolled in the study but did not receive any study treatment.
Arm/Group | MDS or CMML: IV Decitabine | MDS or CMML: ASTX727 | MDS or CMML: Not Treated | AML: IV Decitabine | AML: ASTX727 | AML: Not Treated
All-Cause Mortality (participants affected / at risk) | 2/132 | 56/130 | 0/5 | 5/78 | 61/80 | 2/2
Serious Adverse Events (participants affected / at risk) | 24/132 | 81/130 | 0/5 | 19/78 | 65/80 | 1/2
Other Adverse Events (participants affected / at risk) | 127/132 | 130/130 | 0/5 | 70/78 | 76/80 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDS or CMML: IV Decitabine (N=132) | MDS or CMML: ASTX727 (N=130) | MDS or CMML: Not Treated (N=5) | AML: IV Decitabine (N=78) | AML: ASTX727 (N=80) | AML: Not Treated (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 33 | 0 | 4 | 21 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2 | 0
Proctitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 1 | 2 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Polyserositis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sudden Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 6 | 17 | 0 | 4 | 16 | 0
Sepsis (Infections and infestations) | 0 | 10 | 0 | 0 | 3 | 0
Cellulitis (Infections and infestations) | 2 | 5 | 0 | 1 | 4 | 0
Diverticulitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peritonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 5 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis Aspergillus (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Exposure To Communicable Disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Extravasation Blood (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Loss Of Personal Independence In Daily Activities (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDS or CMML: IV Decitabine (N=132) | MDS or CMML: ASTX727 (N=130) | MDS or CMML: Not Treated (N=5) | AML: IV Decitabine (N=78) | AML: ASTX727 (N=80) | AML: Not Treated (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 90 | 0 | 30 | 47 | 0
Neutropenia (Blood and lymphatic system disorders) | 45 | 79 | 0 | 8 | 27 | 0
Anaemia (Blood and lymphatic system disorders) | 47 | 72 | 0 | 21 | 41 | 0
Leukopenia (Blood and lymphatic system disorders) | 23 | 37 | 0 | 4 | 9 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 8 | 0 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 7 | 0 | 1 | 7 | 0
Conjunctival Haemorrhage (Eye disorders) | 1 | 7 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 26 | 64 | 0 | 8 | 15 | 0
Nausea (Gastrointestinal disorders) | 23 | 63 | 0 | 4 | 17 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 54 | 0 | 1 | 17 | 0
Vomiting (Gastrointestinal disorders) | 4 | 26 | 0 | 3 | 10 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 23 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 20 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 9 | 0 | 0 | 6 | 0
Toothache (Gastrointestinal disorders) | 2 | 9 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 8 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 23 | 68 | 0 | 2 | 9 | 0
Oedema Peripheral (General disorders) | 10 | 36 | 0 | 8 | 16 | 0
Asthenia (General disorders) | 6 | 29 | 0 | 6 | 20 | 0
Pyrexia (General disorders) | 10 | 27 | 0 | 6 | 18 | 0
Chills (General disorders) | 2 | 13 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 9 | 0 | 0 | 0 | 0
Pain (General disorders) | 5 | 8 | 0 | 2 | 4 | 0
Peripheral Swelling (General disorders) | 2 | 7 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 16 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 16 | 0 | 1 | 8 | 0
Cellulitis (Infections and infestations) | 1 | 11 | 0 | 2 | 6 | 0
Nasopharyngitis (Infections and infestations) | 1 | 10 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 10 | 0 | 1 | 6 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 24 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 16 | 0 | 4 | 8 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 7 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 20 | 0 | 1 | 6 | 0
Blood Creatinine Increased (Investigations) | 4 | 17 | 0 | 1 | 6 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 14 | 0 | 1 | 5 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 4 | 11 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 3 | 10 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 3 | 10 | 0 | 3 | 4 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 3 | 7 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 43 | 0 | 5 | 12 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 27 | 0 | 4 | 15 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 14 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 14 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 12 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 9 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 9 | 0 | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 7 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 32 | 0 | 2 | 8 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 26 | 0 | 4 | 9 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 21 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 18 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 13 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 11 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 19 | 50 | 0 | 2 | 6 | 0
Dizziness (Nervous system disorders) | 13 | 42 | 0 | 2 | 8 | 0
Insomnia (Psychiatric disorders) | 3 | 19 | 0 | 4 | 9 | 0
Anxiety (Psychiatric disorders) | 4 | 10 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 10 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 10 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 7 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 45 | 0 | 3 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 40 | 0 | 2 | 9 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 26 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 16 | 0 | 2 | 7 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 15 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 6 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 | 17 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 16 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 13 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 12 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9 | 0 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 8 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 7 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 6 | 16 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 10 | 0 | 3 | 8 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 3 | 9 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 4 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 0
Tongue Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 2 | 4 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 2 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03306264/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (for MDS and CMML) (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT03306264/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (for AML) (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03306264/SAP_002.pdf